CLINICAL TRIAL: NCT07086404
Title: Early Exploratory Clinical Study of GC012F Injection in Refractory Idiopathic Inflammatory Myopathy
Brief Title: GC012F Injection in Refractory Idiopathic Inflammatory Myopathy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daishi Tian (Other)
Collaborators: AstraZeneca Global R&D (China) Co., Ltd. (Unknown); Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Daishi Tian, Chief Physician of Neurology, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC012F in IIM
Record Dates: First submitted 2025-07-07; First posted 2025-07-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Inflammatory Myopathy (IIM)
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3.0×10^5 CAR-T cells/kg (Experimental)
  Interventions: Drug: GC012F Injection infusion

INTERVENTIONS:
Drug: GC012F Injection infusion — GC012F Injection infusion will be performed within 48-72 hours after the end of lymphodepleting preconditioning.

SUMMARY:
This is a single-arm, open-label, early exploratory clinical study to evaluate the safety and efficacy of GC012F Injection in subjects with refractory idiopathic inflammatory myopathy and to assess the pharmacokinetic and pharmacodynamic profiles.

This study consists of screening period, apheresis period, baseline period, lymphodepleting preconditioning period, pre-infusion evaluation period, CAR-T cell infusion period and follow-up period.

Eligible subjects will undergo apheresis and receive infusion following the manufacture of the CAR-T product. Subjects will receive lymphodepleting preconditioning before CAR-T cell infusion and will be assessed before infusion. If the criteria for cell infusion are met, CAR-T cell infusion will be performed and the infusion dose in the same group or subsequent treatment groups may be adjusted according to the safety and clinical response.

A total of 1 dose group will be set for CAR-T cell infusion dose in this study: 3 × 10^5/kg. Approximately 12 subjects are planned to be enrolled. Subjects will be monitored for dose-limiting toxicity (DLT) within 28 days following the infusion of GC012F Injection. For the first 3 patients receiving infusions of GC012F, 3 additional patients will be included in this cohort if no more than 1/3 of the patients experience DLTs at a given dose level. If 2/3 or more DLTs occur at this dose level, a spare dose of 2.0 × 10^5/kg or 1.0 × 10^5/kg may be administered to subsequent subjects following discussion between the investigator and the partner. If no more than 1 out of the first 6 subjects experiences a DLT, 6 additional subjects will be enrolled. Once 2 subjects experience DLTs, the investigator and the partner will discuss and decide whether to use a spare dose group of 2.0×10^5/kg or 1.0×10^5/kg.

After the first 3 subjects have all completed the 28-day DLT observation period, the Safety Monitoring Committee (SMC) will conduct an assessment based on clinical safety and pharmacokinetic data (if available). Subsequently, the SMC may, depending on the safety profile and study progress, request an increased frequency of safety committee assessments and reviews. After completing the DLT observation period for all subjects in this dose group, all clinical study data collected during the DLT observation period for this dose group, especially safety data, will be assessed, and whether to add new subjects to this dose group and whether to explore a different dose group will be decided upon discussion between the investigator and the partner.

Following CAR-T cell infusion, subjects will be followed for safety, cell proliferation and survival, and efficacy until the subject withdraws from the study and refuses subsequent follow-up, or dies, or withdraws consent, or is lost to follow-up, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 1) The subject or his/her legally acceptable representative voluntarily signs the written informed consent form and is willing and able to comply with the procedures of this study; 2) Aged 18 to 70 years (inclusive) at the time of signing informed consent, male or female; 3) Patients should meet the following criteria:

  1. Subjects with suspected or confirmed idiopathic inflammatory myopathy (IIM) based on the 2017 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria and at least one proximal limb muscle strength of less than or equal to Grade 4; patients with immune-mediated necrotizing myopathy (IMNM) may be included if he/she meets other inclusion criteria and does not meet all exclusion criteria and the investigator assesses that the patient has no safety instability;
  2. Active myositis on muscle biopsy or muscle magnetic resonance imaging (MRI) within the screening period or within 6 months prior to screening;
  3. Positive (+ or above) for at least one myositis-specific antibody (MSA) or myositis-associated antibody (MAA) (including anti-TIF-1γ, NXP-2, Mi-2α, Mi-2β, MDA-5, SAE-1/2, SRP, HMGCR, Jo-1, PL-7, PL-12, HA, EJ, OJ, KS, Zo, PM-Scl100, PM-Scl75, SSA/Ro-52, SSB/LA, Ku, RNA-PIII, cN1A, etc.);
  4. At screening, the subject must have moderate to severe IIM, defined as manual muscle testing (MMT) < 142 and 2 of the following criteria are met:

     * PGA (VAS) ≥ 2 cm (VAS 10 cm scale);
     * PtGA (VAS) ≥ 2 cm (VAS 10 cm scale);
     * Health assessment questionnaire (HAQ) > 0.25;
     * Increase in one or more muscle enzymes (CK, LDH, AST, ALT) is ≥ 1.5 × ULN;
     * Extramuscular global assessment (Myositis Disease Activity Assessment Tool [MDAAT]) ≥ 2.0 cm (VAS 10 cm scale); 4) Muscle enzyme increased (CK) ≥ 2 × ULN; 5) Inadequate response or intolerance to corticosteroids and at least 2 immunosuppressants and/or biologic agents; 6) If the patient is taking corticosteroids, the dose of prednisone should not exceed 40 mg/day (or equivalent dose of other corticosteroids) within 3 weeks before apheresis, and the dose is not uptitrated within 3 weeks before apheresis and not changed within 4 weeks before infusion (Note: under the premise that the subject's disease under study is controlled, the investigator may consider reducing the dose of corticosteroids before apheresis, lymphodepletion, and infusion); 7) Life expectancy ≥3 months; 8) Laboratory test results must meet the following criteria at screening (except for those related to the corresponding disease under study):

  <!-- -->

  1. Neutrophil count > 1.0 × 10^9/L, Hemoglobin ≥ 80g/L, platelet count ≥ 50 × 10^9/L;
  2. Alanine aminotransferase ≤ 3 × upper limit of normal (ULN); aspartate aminotransferase ≤ 3 × ULN (unless the increases in alanine aminotransferase and/or aspartate aminotransferase are assessed by the investigator as related to polymyositis [PM] or dermatomyositis [DM]); total bilirubin (TBIL) < 2 × ULN (direct bilirubin [DBIL] ≤ 1.5 × ULN for subjects with Gilbert's syndrome);
  3. Creatinine clearance ≥ 60 ml/min;
  4. Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN;
  5. Left ventricular ejection fraction (LVEF) ≥ 50% as diagnosed by echocardiogram, with no evidence of pericardial effusion as determined; 9) Women of childbearing potential must:

  <!-- -->

  1. Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result at screening as confirmed by the investigator;
  2. Agree to avoid breastfeeding during the study period and until at least 2 years after infusion of GC012F Injection, or until two consecutive flow cytometry tests indicate that CAR-T cells are no longer present (whichever occurs later); 10) Male subjects with sexual partners and female subjects of childbearing potential must agree to use highly effective contraception methods (e.g., oral contraceptives, intrauterine devices, or condoms) starting from screening and continuing for at least 2 years after GC012F Injection infusion or until two consecutive flow cytometry tests indicate that CAR-T cells are no longer present (whichever occurs later). Male subjects must agree to use condoms during any sexual contact with pregnant women or women of childbearing potential for at least 2 years after GC012F Injection infusion, even if they have undergone successful vasoligation.

     11) The required venous access for collection can be set up, with no contraindications for leukapheresis.

     Exclusion Criteria:
* 1) Documented inclusion body myositis (IBM), drug-induced PM or DM, tumor-related PM or DM, amyopathic DM, non-inflammatory myopathy (e.g., muscular dystrophy); for patients with PM or DM, they were > 40 years of age at onset of PM or DM symptoms and the diagnosis time is less than 3 years, and the investigator considered a possible malignancy based on the patient's clinical presentation; 2) Uncontrolled extramuscular disease impairment associated with PM or DM:

  1. Interstitial lung disease (ILD): Forced vital capacity (FVC) < 55% or requiring oxygen therapy;
  2. Severe dysphagia manifestations, that will increase the risk associated with the patient's participation in the clinical trial, as judged by the investigator;
  3. Severe cardiac manifestations (e.g., congestive heart failure, arrhythmia, conduction abnormality requiring treatment or myocardial infarction) that, in the judgment of the investigator, will increase the risk associated with the patient's participation in the clinical trial; 3) Patients with severe muscle injury who meet one of the following criteria:

  <!-- -->

  1. Myositis damage index (MDI) ≥ 5;
  2. Severe proximal muscle atrophy of the upper or lower extremities as shown on MRI;
  3. Severe proximal muscle atrophy of the upper or lower extremities as found by clinical examinations; 4) History of severe hypersensitivity or allergy; 5) Contraindications or hypersensitivity to fludarabine, cyclophosphamide, or any component of the investigational product; 6) Presence of the following cardiac disorders:

  <!-- -->

  1. New York Heart Association (NYHA) Class III or IV congestive heart failure;
  2. Myocardial infarction or coronary artery bypass grafting within 6 months prior to screening;
  3. History of clinically significant ventricular arrhythmia or unexplained syncope not due to a vasovagal reaction or dehydration, or QTc interval > 480 milliseconds at screening;
  4. History of severe non-ischemic cardiomyopathy; 7) Any active malignancy or history of malignancy within 5 years prior to screening. Exceptions include curatively treated early stage tumors (carcinoma in situ or stage I tumors, non-ulcerative primary melanoma with a depth of less than 1 mm and no involvement of lymph nodes), cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, in-situ carcinoma of cervix, or in-situ carcinoma of breast that has been potentially curatively treated; 8) Clinically significant hemorrhage symptoms or a definite tendency to hemorrhage within 6 months prior to screening, such as hemorrhage of digestive tract and hemorrhagic gastric ulcer; hereditary or acquired hemorrhage or thrombotic tendencies (e.g., hemophilia, coagulation disorders, and hypersplenism); arterial or venous thrombotic events within 6 months prior to screening, such as cerebrovascular diseases (including cerebral hemorrhage and cerebral infarction), deep vein thrombosis and/or pulmonary embolism; 9) Severe underlying medical conditions such as:

  <!-- -->

  1. Evidence of viral, bacterial, fungal, or other infections that are uncontrolled or need systemic intravenous treatment;
  2. Clear clinical evidence of dementia or altered mental status;
  3. Any other central nervous system disease or history of neurodegenerative diseases, such as epilepsy, seizure, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, and psychosis; 10) Any of the following test results is positive:

  <!-- -->

  1. Human immunodeficiency virus (HIV) antibody positive;
  2. Hepatitis B surface antigen (HBsAg) positive; or hepatitis B core antibody (HBcAb) positive, and hepatitis B virus (HBV) -DNA above the lower limit of detection of the assay;
  3. Hepatitis C virus (HCV) antibody positive and HCV RNA above the lower limit of detection of the assay;
  4. Syphilis antibody positive; 11) Active tuberculosis or latent tuberculosis that has not been treated appropriately prior to screening; 12) Receipt of other investigational products within 4 weeks prior to signing the ICF, or if the time from the last dose of a previous investigational product to the ICF signing date is still within 5 half-lives of that drug (whichever is longer); 13) Thymectomy within 12 months prior to signing the ICF; 14) Receipt of drugs targeting B cells within 3 months prior to signing of the ICF; 15) Receipt of other biologic agents within 3 weeks prior to apheresis or within 8 weeks prior to infusion; 16) Major surgery within 8 weeks prior to signing the ICF, or planned surgery during the study; 17) History of organ transplantation; 18) Prior therapy targeting cluster of CD19 and/or BCMA-targeted therapy, or CAR-T product therapy targeting any antigen; 19) Pregnant women, breastfeeding women who do not agree to discontinue breastfeeding, or males and females who plan to conceive during the study or within 1 years after receiving study treatment; 20) Any condition, as determined by the investigator, that would interfere with the subject's full participation in the study, confound the study results, or render participation in the study not in the best interest of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with dose-limiting toxicity (DLT) within 28 days after infusion. | Within 28 days after infusion.
Post-infusion adverse events (AEs) and their proportion. | Within 672 days (96 weeks) after infusion.

SECONDARY OUTCOMES:
CAR-T cell count in peripheral blood at each time point. | Within 672 days (96 weeks) after infusion.
Quantification of cytokines in peripheral blood at each time point. | Within 672 days (96 weeks) after infusion.
CAR transgene copy number in peripheral blood at each time point. | Within 672 days (96 weeks) after infusion.
Quantification of immunoglobulins in peripheral blood at each time point. | Within 672 days (96 weeks) after infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical Colledge, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No